CLINICAL TRIAL: NCT00942110
Title: Examination of Association Between Glucose, Lipid Metabolism and Obstructive Sleep Apnea
Brief Title: Alterations in Postprandial Glucose and Lipid Metabolism in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Toru Oga, Medical doctor, Kyoto University, Graduate School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-311
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Postprandial glucose, lipid metabolism; humoral factors
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPAP (Experimental)
  Interventions: Device: CPAP treatment

INTERVENTIONS:
Device: CPAP treatment — maintains upper airway patency and minimizes the obstructive events
  Other Names: REMstar (Respironics), Auto Set(Resmed), Goodnight (Tyco Healthcare)

SUMMARY:
The purpose of this study is to examine postprandial glucose and lipid metabolism in patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is an increasingly prevalent condition that is characterized by repetitive upper airway obstructions. OSA has been independently associated with insulin resistance, suggesting that OSA may contribute to the development of type 2 diabetes and the metabolic syndrome. Recently, postprandial glucose and lipid have been reported as excellent predictors for mortality and cardiovascular risk. However, the association between postprandial glucose, lipid metabolism and OSA are not clear. In addition, humoral factors such as ghrelin and leptin are associated with obesity and OSA, but postprandial changes of which in patients with OSA are not well known. The aim of present study is to examine postprandial glucose and lipid metabolism, humoral factors in OSA before and after 3 months of continuous positive airway pressure (CPAP) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects on admission for sleep study under the Respiratory Care and Sleep Control Medicine, Kyoto University Hospital.
* Subjects diagnosed with OSA (apnea hypopnea index >=5/hour) by overnight polysomnography.

Exclusion Criteria:

* Subjects treating for acute infections or malignancy.
* Subjects with severe anemia, diabetes,and renal failure.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
postprandial metabolic markers including glucose, cholesterol, triglyceride, ghrelin, leptin | baseline and 3 months after CPAP

SECONDARY OUTCOMES:
respiratory events (ie. apnea-hypopnea index) | baseline and 3 months after CPAP
inflammatory biomarkers (ie. IL-6, CRP) | baseline and 3 months after CPAP
quality of life | baseline and 3 months after CPAP
sleep quality | baseline and 3 months after CPAP
sympathetic activity in urine | baseline and 3 months after CPAP
appetite | baseline and 3 months after CPAP
endothelial function | baseline and 3months after CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Chin, MD,PhD, Principal Investigator — Kyoto University, Graduate School of Medicine; Yuichi Chihara, MD,PhD, Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University Graduate School of Medicine, Kyoto, Kyoto, Japan